CLINICAL TRIAL: NCT02340858
Title: Safety and Efficacy of Irreversible Electroporation (IRE) for Breast Cancer
Brief Title: Percutaneous Irreversible Electroportion for Unresectable Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JF-20150112(3)
Record Dates: First submitted 2015-01-12; First posted 2015-01-19 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2019-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NanoKnife LEDC System (Experimental): 90 pulses of 70 microseconds each in duration will be administered per electrode pair.
  Interventions: Device: NanoKnife LEDC System
- Control (No Intervention): The patients without treatment

INTERVENTIONS:
Device: NanoKnife LEDC System — Irreversible electroporation (IRE) is a method to induce irreversible disruption of cell membrane integrity (loss of cell homeostasis) resulting in cell death without the need for additional pharmacological injury. Because IRE is a non-thermal technique, changes associated with perfusion-mediated tissue cooling (or heating) are not relevant. While cells in the ablation region are destroyed, the underlying extracellular matrix is not damaged thus allowing tissues in the ablation zone to heal normally.
  Other Names: NanoKnife
  Arms: NanoKnife LEDC System

SUMMARY:
This trial is studying how well Irreversible Electroportion (IRE) therapy works in treating patients with breast cancer. IRE kills tumor cells by Electrical impulses creating nano-pore on the cell membrane and inducing target cell death.This may be an effective treatment for patients with unresectable breast cancer.

DETAILED DESCRIPTION:
This is a phase I/II non-randomized exploratory study. All fully eligible and registered patients will undergo imaging by mammography, ultrasound, and breast MRI. The primary and secondary objectives of the study are described below.

OBJECTIVES

Primary

Treatment efficacy as measured by modified Response Evaluation Criteria In Solid Tumors (RECIST) criteria by Computed Tomography (CT) or Magnetic Resonance (MR) imaging.

secondary

Safety using Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 criteria.

To describe the adverse events associated with IRE To prospectively gather pain assessment data on cryoablation and surgical resection Explore technical variables that may affect the success of IRE

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years or older with unresectable breast cancer, not amenable/willing to adenomammectomy.
2. breast carcinoma diagnosed by core needle biopsy.
3. Any menopausal status.
4. No history of en bloc open surgical biopsy and/or lumpectomy for diagnostic/treatment of the index breast cancer.
5. Tumor size ≤ 5.0 cm in greatest diameter. Largest size measured by required scans (mammogram, ultrasound and MRI) will be used to determine eligibility.
6. Tumor enhancement on pre-study MRI.
7. Tumor with < 25% intraductal components in the aggregate.
8. Progressed within 12 months from prior adjuvant or progressed within 1 month from prior advanced/metastatic endocrine breast cancer therapy,
9. Non-pregnant and non-lactating. Patients of childbearing potential must have a negative serum or urine pregnancy test.
10. Adequate breast size for safe IRE. Male breast cancer patients and female breast cancer patients with breasts too small to allow safe IRE are not eligible as the minimal thickness of the breast tissue does not lend itself to IRE. NOTE: For patients with breast implants, the treating physician must document that adequate distance exists between the lesion and the implant to ensure that the ablated lesion will not contact or jeopardize the implant.
11. Adequate organ and marrow function, resolution of all toxic effects of prior therapy or surgical procedures
12. Patient must agree to provide tumor tissue from metastatic tissue at baseline.

Exclusion Criteria:

1. Patients with multifocal and/or multicentric ipsilateral breast cancer, multifocal calcifications, or evidence of excessive DCIS.
2. History of rotational vacuum assisted core biopsies, en bloc open surgical biopsy and/or lumpectomy for diagnosis/treatment of the index breast cancer.
3. Prior or planned neoadjuvant chemotherapy for breast cancer.
4. Patients with thrombocytopenia and or any other coagulation abnormality

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Treatment efficacy as measured by modified Response Evaluation Criteria In Solid Tumors (RECIST) criteria by Computed Tomography (CT) or Magnetic Resonance (MR) imaging. | 3 months post treatment to 24 months

SECONDARY OUTCOMES:
Safety using Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 criteria. | 1 day post treatment to 3 weeks

OTHER OUTCOMES:
Adverse Events | 1 day post surgery to 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lizhi l Niu, Study Director — FUDA Cancer Hospital
Locations (1):
- FUDA Cancer Hospital, Guangzhou, Guangdong, China